CLINICAL TRIAL: NCT03768115
Title: Use of Autologous Plasma Eyedrops Therapy for Severe Dry Eye in Singapore
Brief Title: Autologous Plasma Treatment for Severe Dry Eye Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The inclusion criteria for plasmapheresis is too stringent to get any potential subjects.
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Health Science Authority Singapore (Unknown)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R945/54/2012; 2018/2855 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Autologous crimped plasma segments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Autologous Plasma Eye Drop — Autologous plasma crimped segments

SUMMARY:
Patients with severe dry eye who have exhausted conventional treatment are not uncommon and are difficult to manage. They and their physicians are helpless when faced with these scenarios. A small HPRG group, Health Science Authority (HSA) and IRB approved study of autologous plasma eye drop therapy for patients with recalcitrant dry eye has been completed recently by investigators at the Singapore National Eye Centre. The unique feature of the previous protocol was that the autologous plasma preparation was made and contained in sealed segments of intravenous tubing until use by the patient. The study showed that the corneal fluorescein staining of patients who regularly used autologous plasma over a 6 week period improved significantly. Additionally, there was a significant reduction in the total number of topical eye drop treatment required. Investigator did not encounter any cases of infected eye drop preparation or any cases of eye infection. Seventy percent of these patients would recommend this treatment to their relatives and friends suggesting that this form of treatment is a valuable additional modality for dry eyes. Now, investigator would like to extend the short-term pilot study into a long-term single arm clinical trial, in order to determine the best protocol/logistic for this treatment that is practical and still effective, and allowing for more than one plasmapheresis during the study. To achieve this, investigator aim to perform a longitudinal prospective study of patients with severe dry eye who cannot be satisfactorily managed with conventional dry eye treatments using a proposed regime for plasmapheresis and plasma storage.

DETAILED DESCRIPTION:
Dry eye is a multi-factorial disease that is frequently encountered in ophthalmological practice. Common dry eye symptoms include eye irritation, heaviness of the eyelids, blurred vision and light sensitivity. The worldwide prevalence of dry eye is generally high. In Asia, dry eye may affect up to 22% of adults above 40 years in China and Japan. In Asian patients older than 65 years, prevalence rates of dry eye can be as high as 80% if diagnosis is based on abnormal tear stability, or as high as 60% on meibomian gland dysfunction (MGD), a major cause of tear instability.

In a Singapore study, dry eye significantly impacted the quality of life of patients as a consequence of constant interference with daily activities, such as navigating stairs, recognizing friends or watching TV. Additionally, patients with severe dry eye reported that this condition is comparable to dialysis or severe angina, which emphasizes the enormous impact the dry eye disease has on patients.

Dry eye disease presents a significant socio-economic problem. The overall economic burden of dry eye management and treatment has been reported to be US$ 3.84 billion per annum in the American healthcare system and up to US$ 1.1 million per thousand persons per annum in Europe. The economic cost of dry eye is also high in Singapore. In 2009, the Singapore National Eye Centre (SNEC) treated 54,051 dry eye patients and the corresponding total cost for medication amounted to SG$ 181,354 in this single centre (unpublished data). This data does not account for other over-the-counter lubricants that were purchased by dry eye patients at pharmacies outside SNEC, so the cost may even be significantly higher.

Most dry eye patients can be successfully managed with lubricants, punctal occlusion, steroid and/or cyclosporine eye drops. However, some patients with severe dry eye and likely underlying diseases (for example graft versus host disease, rheumatoid arthritis and Sjögrens-Syndrome), who have exhausted conventional treatments may amount to 10-20 cases a year and are difficult to manage. These patients and their physicians are helpless when faced with these scenarios. These patients have attempted different kinds of eyedrops such as longer acting gels, doxycycline, punctal plugs, cyclosporine and even topical steroids. Many of these patient's epitheliopathy, vision, and tear function are at best, stable at a very unsatisfactory level. Furthermore, all of these patients are currently using eyedrops to the frequency of half hourly to hourly, and this further affects work productivity and quality of life. The situation is so critical in these patients that should a form of therapy be available that can improve the quality of life, such as reducing the number of eyedrops required per day, it would constitute a definite advance, even if the disease cannot be reversed, or vision not clearly improved.

A small HPRG group, HSA and IRB approved study of autologous plasma eye drop therapy for patients with recalcitrant dry eye has been completed by investigators at the Singapore National Eye Centre (SNEC). The IRB approval no was 2010/137/A dated 12. April 2010. The HSA CTC approval no was CTC 1000230 dated 22/06/2010. Briefly, the unique feature of the previous protocol was that the autologous plasma preparation was made and contained in sealed segments of intravenous tubing until use by the patient. The study showed that the corneal fluorescein staining of patients who regularly used autologous plasma over a 6-week period improved significantly. Additionally, there was a significant reduction in the total number of topical eye drop treatment required. Investigator did not encounter any cases of infected eye drop preparation or any cases of eye infection. Seventy percent of these patients would recommend this treatment to their relatives suggesting that this form of treatment is a valuable additional modality for dry eyes. In addition to these quantitative outcomes, believe that there are some patients with particularly remarkable results that cannot be quantified easily. For example, one patient, having had years of unsuccessful treatment with various formulations, claimed that 'this is the only type of eyedrops that make any difference'. The scientific evidence for the use of full strength plasma is further strengthened by a recently published study that showed superiority of undiluted serum over half strength serum in relieving symptoms of dry eye and epithelial damage.

What would be the next step for the evaluation of autologous plasma treatment in severe dry eye? This form of treatment in severe dry eye is not appropriate for a randomised controlled study for the following reasons: First, two randomised studies have shown the efficacy of autologous serum compared to 'standard therapy, reported in 2004 and 2005. For a proposed randomised study to be ethical, there has to be equipoise. In this situation, having a control group of say 'saline' in crimped tubings is not ethical for severe dry eye. Second, there is no comparison treatment that is available in the Singapore context. The internationally accepted treatments for severe/recalcitrant dry eye are tarsorrhaphy, prosthetic replacement of ocular surface ecosystems (PROSE) and autologous serum/plasma. The PROSE is a form of sclera contact lens that is not available in Singapore and is very expensive (US$3000-5000). Tarsorrhaphy is a form of surgery (invasive treatment) and is obviously not suitable for many cases of bilateral severe dry eyes, since closing the eyelids will prevent proper vision, in addition to cosmetic blemishes. Third, all of the current severe dry eye patients are using different lubricant formulations up to half hourly, many of these formulations such as Systane Ultra gels are much more effective than saline. These patients are constantly requesting for more effective solutions and are understandably unwilling to use additional saline eyedrops as part of the comparison group, if they are not randomised to receive autologous plasma. In any arm of a study on severe dry eye, the study intervention is in addition to the existing treatment (lubricants, doxycycline etc). The one major reason for decreased quality of life is the requirement for very frequent eyedrops, it is not surprising that willingness to use yet another eyedrop that is less effective than their current existing drops is low. Therefore, an attempt to do a randomised study that requires saline in one arm on such patients will be doomed to fail due to lack of cooperation. Masking of treatment status is not possible since the control patients would be aware that they did not have plasmapheresis. The only possibility to do a randomised study will be in moderate dry eye (rather than severe recalcitrant ones). However, this is not currently the priority at Singapore National Eye Centre, where the immediate concern is to address the patients' unmet needs, and the patients with moderate dry eye, unlike their severe counterparts, have several viable alternatives in the treatment repertoire.

If the most suitable methodology is a single arm prospective study, their outcomes can still be compared to other severe dry eye patients who for some reason, did not want to participate. In the current scenario, where there is no real alternative strategy for treatment of severe dry eye, autologous plasma should be definitely used and evaluated further. If the regulatory bodies approved this, it would be unethical not to consider this, since autologous plasma has been shown to be safe and effective in the short term. Some desperate severe dry eye patients have considered alternative ways of obtaining the autologous serum, for example, from private clinics and from neighbouring countries. These treatments may be obtained at much lower costs compared to plasmapheresis, but not necessarily safer, outside the context of a clinical study. In my opinion, based on managing these cases over the last 6 years, the relevant question is not whether autologous plasma should be used, but rather, how such therapy can be used in a protocol that is practical, convenient and acceptable.

In the above pilot study, the plasma eye drops were prepared at the hematology centre at SGH. After the completion of the study, investigator has been informed by the hematology centre that their new accreditation status will prohibit preparation of autologous plasma segments by crimping within the premises even though they can still perform the plasmapheresis. This increases the inconvenience of the whole dispensing procedure and may increase the non-refrigerated time of the harvested plasma. In addition overseas experience, for example, at the Methodist Hospital in Houston Texas show that it is safer and more efficient for blood professionals to handle blood products for clinical use rather than other types of health professionals. For this reason investigator seek the assistance of blood group services at HSA to perform this part of the study. The facility at HSA has the ability to perform crimping of the intravenous tube, so it may not be necessary to use the current multi-head crimper. The current crimper is nevertheless, available for use if desired. A further enhancement of the procedure can be performed at HSA, using a sealing process that connects contiguous intravenous tubes without using 3 way taps. This will ensure an entirely closed environment where the plasma is not exposed to the environment until just before using the eyedrop.

As autologous plasma treatment is currently advocated in our centre only for severe/recalcitrant dry eye, it is not expected that the costs of such therapy can be lowered significantly from the scale of the service since patient number is small at any one time. Investigator expects that only about 10-20 such patients may appear per year, but these account for a considerable number of hospital visits per year. The main problem with autologous plasma as a treatment modality is the one-time cost associated with the plasmapheresis itself. In order to make the costs of autologous plasma more realistic and affordable, investigator would like to explore the storage of plasma for a longer time than 6 weeks or 3 months from a single plasmapheresis. As conditions (temperature and hygiene) of plasma storage is much more predictable at a central storage facility at HSA, investigator will explore storing half of the extract patient's plasma and dispensing it after the exhaustion of the initial supply, without necessitating further plasmapheresis and incurring additional costs.

Many of the dry eye patients use Restasis (topical cyclosporine 0.05% emulsion) which costs S$70 every three weeks on a long term basis. In the pilot study above, patients on autologous plasma drops were able to cease Restasis during the time when they use the autologous plasma. In other words, over the course of about 21 weeks, a patient who uses Restasis would have a greater expenditure for the medications than a patient who had autologous plasma drops. The autologous plasma user may also save additionally from the reduced number of eyedrops used daily, and therefore buying fewer lubricants in 21 weeks. This difference will be even greater since investigator anticipate that a single plasmapheresis can produce sufficient eyedrops for a period longer than 21 weeks.

It is believed that plasma eyedrops is superior to conventional eyedrops due to the presence of various anti-inflammatory proteins such as transforming growth factor-beta in plasma. Based on the current literature, it is difficult to ascertain the shelf life of the beneficial proteins after plasma is frozen at -20°C. A pilot study developed a closed, cascade-filtration system that was an effective method for the production of high-quality, low-pyrogen autologous serum. This processing method broadly complied with Food and Drug Administration requirements for reinjection of biological substances. Variable growth factor stability was observed at +4°C and above. Stability of transforming growth factor beta1, substance P, nerve growth factor, calcitonin gene-related peptide, insulin-like growth factor 1, and epidermal growth factor was evaluated at -15°C, +4°C, +25°C, +37°C, and +42°C at different time intervals (hours to weeks). Transforming growth factor beta1, nerve growth factor, epidermal growth factor, and insulin-like growth factor 1 were more temperature and time resistant, but substance P and calcitonin gene-related peptide significantly degraded at +4°C in 24 hours. Endotoxin and lipid peroxidation by-products were not significantly increased by processing.

A very recently published study by a group with much experience in autologous serum treatment for dry eye obtained whole blood from 10 volunteers and prepared 100% (AS100), 50% (AS50), and 20% (AS20) serum eye drops. Epitheliotrophic factors including EGF, fibronectin, vitamins A and E, albumin, and immunoglobulin A were quantified before and after storage for 7 days at 6°C or 3 and 6 months at -20°C. Human corneal epithelial (HCE) cell lines were used to investigate proliferation, migration, and overall wound healing potency of the cells in response to different serum preparations. The proliferation, migration, and wound healing of HCE cells were measured after incubation with different serum eye drop concentrations and after different storage conditions. The results show that the concentration of epidermal growth factor, fibronectin, vitamins A and E, immunoglobulin A, and albumin showed no significant reduction over the test period. Proliferation, migration, and wound healing of HCE cells was significantly better after incubation with undiluted serum in comparison with diluted serum. No significant loss of cytokine concentration, wound healing, and proliferation effect in HCE culture of AS100, AS50, and AS20 could be detected over the 6 months of storage. This study suggests that storing a portion of the autologous plasma in a reliable fashion for 6 months should not result in greatly decreased efficacy for dry eye treatment.

Now, investigator aim to provide an autologous plasma eye drop treatment as a clinical service provided by Singapore National Eye Centre to any patients who cannot be satisfactorily managed with conventional dry eye treatments (lubricants, punctal occlusion, steroid and/or cyclosporine). Specifically, investigator will determine if the significant beneficial effects of autologous plasma treatment obtained at 6 weeks will persist to 12 months, as a way to evaluate if longer term storage of frozen plasma from a single plasmapheresis remains effective. Secondly, to will determine if the effectiveness of this therapy remains at 24 months compared to pre-treatment assessment, and explore whether specific etiologies of dry eye benefit more from this type of treatment.

Clinical importance At the Singapore National Eye Centre, the principal investigator Dr. Tong runs a specialised dry eye service. During his clinical consultations, he encounters patients with severe dry eye who suffer from persistent poor vision. The number of severe dry eye patients is not high but these patients are devastated by the eye condition. This study is important because it addresses aspects of using autologous plasma treatment for severe dry eye, such as feasibility of storing plasma long term in a central freezer, and the data obtained will determine the best method/protocol for administering the only available treatment for severe dry eye locally.

1 HYPOTHESIS AND OBJECTIVES Chronic severe and recalcitrant dry eye form a small group of patients seen at the Singapore National Eye Centre. The symptoms of blurring, decreased comfort and frequent requirement of eye drops result in reduced quality of life. In a longitudinal prospective study, investigator aim to observe the long-term safety and efficacy of autologous plasma eye drop therapy, the only available form of therapy for severe dry eye patients from the Singapore National Eye Centre.

1.1 Hypothesis To evaluate the long-term efficacy, safety and patient acceptability of autologous plasma eye drop therapy using a protocol developed at our centre.

1.2 Primary Objectives

1. To evaluate the difference in number of eye drops used daily and dry eye symptom severity at 6 weeks to 4 months period and subsequent follow up visits at SNEC after commencement of autologous plasma eye drops in patients with severe/recalcitrant dry eye in the dry eye clinic at Singapore National Eye Centre who has failed all other available standard therapy.

   1.3 Secondary Objectives
2. To evaluate the difference in number of eye drops used daily and dry eye symptom severity between the baseline visit and 1 year after the autologous plasma eye drop treatment has stopped.
3. To explore the treatment outcome in terms of the etiological subtype of the patients (eg., graft versus host, rheumatoid arthritis, etc) to see if particular subgroups respond particularly well to this form of treatment.

1.4 Potential Risks and Benefits: 1.4.1 Potential Risks A possible adverse reaction is the presence of increased redness of the eye and/or increased irritation after commencement of the treatment. This may or may not be due to contamination and subsequent infection of the ocular surface. The signs and symptoms will be managed according to clinical findings. In order to avoid serious infections, especially corneal keratitis, investigator will not include patients with high risks for infection in this study, such as those patients with a persistent epithelial defect, wearing of contact lenses, previous ocular surgery such as penetrating keratoplasty or any other ocular surgery. All adverse reactions will be reported to the IRB. If eye drop contamination is suspected, eye drops will be sent for microbiology, in addition to patient swabs or scrapes sent for microbiology.

Another potential problem during plasmapheresis will be headaches, nausea, transient lowering of blood pressure, tinglings of lips and finger tips, shivers, cramps. Others include, bruising and bleeding from venepuncture site, rarely transient fits, nerve injury or arterial puncture.

1.4.2 Potential Benefits Subjects can undergo autologous plasma eye drops treatment for their dry eye condition.

2 STUDY POPULATION 2.1 List The Number and Nature of Subjects to be Enrolled The number of subjects will be dependent on the number of patients from SNEC who requires this treatment as determined by the physician. This is expected to be not more than 10-20 per year. This amounts to not more than a maximum of 40 patients over 2 years of recruitment.

Attending doctors at Singapore National Eye Centre will determine if treatment is necessary for patients. Informed written consent will be obtained from all participants.

2.5 Subject Replacement Subjects who have dropped out will not be replaced. 3 STUDY DESIGN To evaluate the long-term efficacy, safety and patient acceptability of autologous plasma eye drop therapy using a protocol developed at our centre.

3.1 Study Visits and Procedures 3.1.1 Study Visits and Procedures

1. The study will only include patients who have been referred to the dry eye or cornea clinic at SNEC and only patients found to be suitable will be recruited into the trial.
2. The clinical indications for starting treatment and follow up visits will be at the discretion of the principle investigator but the data obtained on designated study visits will be collected on study case report forms and data entered electronically into a database for analysis. The eligibility will adhere as much as possible to the inclusion criteria in the previous study. However, patients with previous plasmapheresis and autologous plasma treatment (as long as it did not occur within the last 2 weeks) will now be permitted to participate in this study. To address the first aim of the study, the symptoms at one year after the patient stopped the autologous plasma treatment will be compared to that at first follow up visit (6 weeks to 4 months) after commencement of autologous plasma The patients will be permitted to have a repeat plasmapheresis after the first one if the patient opts to do that and a second plasmapheresis deemed indicated by the PI. The duration of treatment from one plasmapheresis will be longer than the 6 weeks in the previous study as more plasma will be extracted and half the plasma volume will be stored for later dispensing (described in detail below). In addition, investigator expect that there may be individual factors which make continued plasma treatment unnecessary. The extent of inflammation may wax and wane in patients with severe dry eye, either as part of the natural history or because of systemic treatment of the condition such as the autoimmune disease. In such cases, the ocular condition may improve after a certain amount of autologous plasma treatment and only require conventional eyedrops subsequently. Therefore, the PI will have the discretion to halt any patient's treatment at any time during the study. Patients are required to pay for the full costs for this clinical service available at SNEC, if they are unwilling to continue with this treatment after the collections from the first plasmapheresis procedures they will be continued to be followed up under this study till 1 year (±6 months) after they stopped using the autologous plasma. The follow up visits for this study is dependent on their SNEC appointments as determined by the PI.
3. From the PI's experience in his clinic, it is expected that less than 10 patients will be recruited in the first year, after careful scrutiny of the presenting clinical features. This study does not require the participants to alter any of their pre-existing dry eye or systemic medications, and will not affect clinical decisions such as insertion of punctal plugs and so on. Surgeries such as cataract surgeries may be performed when indicated at any point in the study. If cataract surgery is necessary, investigator will suspend the autologous plasma treatment for at least one month after surgery. This is not expected to be a frequent occurrence as cataract surgery in the presence of a poor cornea epithelium is unlikely to result in patient satisfaction. The principle investigator may cease the autologous plasma eye drop treatment for any clinical or social reason (for example, if patients do not have further access to a freezer) during the follow up. If this happens, treatment may be re-commenced at any time point by the PI.
4. Beyond the hospital consultation, the patient is required to pay the necessary consumable, , cooler box, plasmapheresis procedures, crimping and storage of autologous plasma, transportation and blood testing charges incurred, which will be made known to the patient. Payment will be made at the SNEC. Patients who meet the criteria outlined in section 'Inclusion Criteria' will undergo plasmapheresis at SGH Hematology Centre. A screening for infectious disease will be conducted. If any of the tests is positive for infectious disease,the patient will not be scheduled for plasmapheresis procedure. The crimping of intravenous tube will be performed by trained personnel at the HSA. Counseling on storage and use of autologous tears will be performed at SNEC.
5. Written informed consent will be obtained from all patients prior any procedure. A standardised documentation of dry eye signs and symptoms will be performed at the baseline visit. It is expected that these patients will be followed up by the PI at the clinically indicated frequency, for example, three monthly, etc. The standardised evaluation form will be implemented during the follow up visits at SNEC when the patient is using autologous plasma treatment until 1 year (±6 months) after they have stopped using autologous plasma treatment and the patient will be considered to have exited the study. However, since dry eye is a chronic disease with possibility of reactivation later, investigator can allow the participant to re-enter the study in subsequent visits if the need arises.

Procedures:

Visit 1 (at SNEC and SGH Hematology Centre):

After written informed consent, patients will be screened for good veins at SGH Hematology Centre. Blood testing at SNEC will be arranged for the patient, preferably on the same day of doctor's consultation or any of the following days. Patients will be screened with the inclusion and exclusion checklist as attached (Appendix A). An appointment for plasmapheresis at SGH Hematology Centre will be scheduled within one month of blood testing. The patient will be counselled on storage and use of autologous tears by trained staff and written instructions are given in the patient information sheet. Baseline parameters will be obtained as in Table 1. Patients with HIV, syphilis, Hepatitis B or Hepatitis C carriers will not be included in the study and their plasmapheresis appointment at SGH Hematogloy Centre will be cancelled. They will no longer be participating in the study.

Visit 2 (at SGH Hematology Centre):

Plasmapheresis be conducted at SGH Hematology Centre. Body temperature, , pulse rate and blood pressure will be assessed at SGH Hematology Centre before the plasmapheresis procedures. A plasma fluid volume of a maximum of 300ml will be collected from patients in a closed bag over a period of up to 60 minutes. The Plasma will be transported to HSA blood services group on the same day for crimping by an experienced technician and storage. Each segment will contain a volume of 150 to 300μl of plasma.

Patients will receive up to half of the crimped plasma segments from courier service, while the other half will be stored in a -80°C freezer at HSA. . When patients have almost completely utilized all the frozen segments, they can contact the SERI coordinator again so that arrangements (date and time) can be made for the second batch to be delivered to them.

Selected subsequents visit (at SNEC) The study outcomes will be assessed as in Table 1. Once patients finished the plasma segments and are keen to continue with the treatment (this occurs any time, they can arrange for the remaining plasma to be delivered to them (without additional plasmapheresis).

If all the autologous plasma has been exhausted: Anytime during the clinical episodes, if the PI finds that continued autologous plasma treatment is indicated and the patient is agreeable, the plasmapheresis can be repeated and the patient will be followed up under this study until 1 years after the autologous plasma treatment has stopped.

Storage of crimped plasma segments by patients:

Patient will be given half of the plasma that was extracted from patient body on the first session. The remaining plasma will be safely stored at HSA in a -80°C freezer. Storage at this central facility is more reliable than at home freezers since such a centralized freezer is not frequently opened and the temperature can be maintained.

Patients will be instructed to store segments in a double zip-lock plastic bag in their household freezer. Every morning, patients defrosted their daily desired number of segments and place them into the fridge at 4°C. Each segment will be opened with alcohol wiped scissors and must be discarded after a single use. Patients will be taught on the opening of segments with alcohol wiped scissors and prescribe small square alcohol swabs from the hospital pharmacy on commencement of the treatment and advice patients on how to obtain further swabs if the supply runs out. Patients are required to use the autologous plasma strictly according to the instructions in the patient information sheet strictly.

Usage:

Patients will use autologous plasma only for application as eye drops. The daily dose is dependent on the patient's requirements. For example, if patients use the plasma 3 times daily, a total of 3 segments should be defrosted each morning. Patients are allowed to continue their existing dry eye medications. However, it is important that the plasma eye drops are instilled at least 5 minutes prior any other eye medications. All existing dry eye medications will be recorded.

The following procedures may be performed:

Difference of Visual Analogue Scale (VAS) for the ocular discomfort between baseline and follow-up visits (continuous variable) A VAS will be applied to evaluate dry eye symptoms as described by Schaumberg et al. (Schaumberg 2007). As shown in Appendix B , the scores will be recorded separately for frequency and severity of dry eye symptoms. The patient will be asked to check a point on a 100-mm line that corresponds to the degree of the symptom. The location of the mark made by the patient for each question will be measured in mm from the left hand side of the 100 mm line and recorded in mm. For the follow up visits, which measured the distance between the mark made by the patient and the central anchor, a negative value will be recorded if left of the anchor and a positive value if right of the anchor.

A global score will be calculated by multiplying the frequency score by the severity score and taking the square root of the result (to transform back to the original scale).

Tear break up time (TBUT) A drop of normal saline will be instilled on a fluorescein strip (Fluorets). The strip will then be introduced into the inferior conjunctival fornix on the right then left eye of the patient.

The patient will blink a few times and close the eyes for few seconds. The patient will be asked to open the eyes, look ahead at the observer's forehead and not blink for as long as possible. The break up time will be defined and recorded as the time between the lid opening and the first appearance of any dry spot on the cornea. The same procedure will be performed on the left eye.

Corneal fluorescein staining score Assessment of positive fluorescein staining will be assessed after recording TBUT. A scoring system will be applied to corneal and conjunctival zones as depicted in Figure 1. Zones with confluent corneal staining and filaments may be documented.

Schirmers I test (Optional) This will be done with the standard strips currently used at SERI (5 mm wide with a notch for folding). No prior anaesthetic will be used. The strips will be positioned over the inferior temporal half of the lower lid margin in both eyes at the same time.

The patient will be asked to close their eyes. Any excessive irritation signs will be noted. The extent of the wetting in each strip will be recorded after 5 minutes of testing, and strips stored at -80˚C until further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dry eye symptoms, who cannot be satisfactorily managed by currently available dry eye medication
2. TBUT ≤10s
3. Presence of corneal fluorescein staining
4. Visual acuity affected by poor tear film quality
5. No contraindication for blood extraction/ plasmapheresis
6. Age between 21 to 99 years old
7. Skin lesions - The skin at the site of venepuncture in the antecubital area should be free of lesions. Donors with boils, open wounds, chronic eczema or any severe skin infection must be rejected.

Exclusion Criteria:

1. Active ocular infection.
2. Any other specified reason as determined by clinical investigator
3. Severe cardiovascular disease
4. Severe respiratory disease
5. Uncontrolled epilepsy
6. Abnormal bleeding conditions
7. Pregnancy
8. Infectious diseases

   * Patients who are known or diagnosed to have HIV, Hepatitis B or Hepatitis C carriers should not be accepted for donation.
   * Patients who have risk factors for infectious diseases should not be accepted for donation.
9. Patients who have been or are being treated for bacteraemia, or have a significant bacterial infection that can be associated with bacteraemia.
10. Unable to come for follow up at the required frequencies and duration. This includes non-Singapore residents who are patients of the dry eye clinic.
11. In order to avoid serious infections, especially corneal keratitis, we will not include patients with high risks for infection in this study, such as those patients with a persistent epithelial defect, wearing of contact lenses, previous ocular surgery such as penetrating keratoplasty or any other ocular surgery.
12. Patients with persistent epithelial defect that requires bandage contact lens

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline dry eye symptoms at 1 year | 1 year
  A Visual Analogue Scale (VAS) will be applied to evaluate dry eye symptoms as described by Schaumberg et al. (Schaumberg 2007). As shown in Appendix B , the scores will be recorded separately for frequency and severity of dry eye symptoms. The patient will be asked to check a point on a 100-mm line that corresponds to the degree of the symptom. The location of the mark made by the patient for each question will be measured in mm from the left hand side of the 100 mm line and recorded in mm. For the follow up visits, which measured the distance between the mark made by the patient and the central anchor, a negative value will be recorded if left of the anchor and a positive value if right of the anchor. The higher the number, implying more symptoms and frequency of experiencing dry eye.
  A global score will be calculated by multiplying the frequency score by the severity score and taking the square root of the result (to transform back to the original scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No